CLINICAL TRIAL: NCT00400673
Title: Two-Step Remission Induction With Risk-Oriented Consolidation (High-Risk: Allogeneic Stem Cell Transplant; Standard-Risk: Multicycle High-Dose Cytarabine With Autologous Blood Stem Cell Support) for Adult Acute Myelogenous Leukemia
Brief Title: A Risk-Oriented Therapeutic Strategy for Adult Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northern Italy Leukemia Group (Other)
Responsible Party: Renato Bassan, MD, Northern Italy Leukemia Group, Ospedali Riuniti, Bergamo (Italy)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NILG-AML 01/00
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Acute myelogenous leukemia; Adult patients; Cytogenetic risk class; Clinico-cytogenetic risk model; Risk-oriented therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy (Other): Risk-oriented chemotherapy for remission induction (application of sequential high-dose cytarabine course to patients unresponsive to standard chemotherapy course 1) and postremission consiolidation(standard risk: blood stem cell supported high-dose cytarabine course [x3]; high risk: allogeneic SCT)
  Interventions: Behavioral: Two-step remission induction and risk-oriented consolidation

INTERVENTIONS:
Behavioral: Two-step remission induction and risk-oriented consolidation

SUMMARY:
The study was set up to assess:

1. A two-step, increasing-intensity remission induction phase. A conventional chemotherapy course (ICE, plus G-CSF) was followed, in unresponsive patients, by sequential high-dose cytarabine (plus G-CSF), aiming to provide an early effective rescue to as many refractory cases as possible.
2. A risk-oriented postremission consolidation phase. The objective was to adopt allogeneic stem cell transplantation (alloSCT) in high-risk (HR) cases, while standard-risk (SR) ones were consolidated with a multicycle high-dose cytarabine-containing program, which included the use of autologous stem cells plus G-CSF to limit drug-related toxicity and intercycle treatment delays.

DETAILED DESCRIPTION:
Adult AML is a difficult-to-treat illness because of both biological and therapeutic reasons.

As to the first point, many patients are aged >50 years and/or present with significant comorbidity and/or AML-related risk features (poor risk cytogenetics, prior myelodysplasia, secondary AML).

As to the second point, standard-type remission induction therapy is ineffective in 20% or more of the patients, whereas the application of the more effective postremission consolidation options (alloSCT, high-dose cytarabine courses) is often flawed by high-grade toxicity which can offset expected benefits, particularly in older age groups (>50-55 years), where therapy-related death rates are seen in 5%-10% of the cases (chemotherapy) or more (transplants).

Against this background an explorative study was developed in which:

1. All patients aged 16-65 years were considered eligible (acute promyelocytic leukemia excluded), including those with an antecedent diagnosis of myelodysplasia/hematological disorder and/or secondary AML. Both age and disease subtype selection criteria are broader than in most studies on adult AML, adhering more closely to the reported epidemiology of the disease.
2. Remission induction was attempted with a two-step regimen, consisting of conventional chemotherapy (ICE: idarubicin/cytarabine/etoposide +G-CSF) followed, only in the case of failure to respond, by a sequential high dose-cytarabine cycle (cytarabine 3 g/m2/bd on days 1,2,8,9; idarubicin on days 3 and 10; G-GSF; cytarabine dosing 2 g/m2 in patients aged >55 years). It was hoped that this choice would optimize salvage rates (hence overall response rates), by allowing more patients (and more fit, uncomplicated ones) to reach the salvage phase, compared to a policy where salvage is usually given after two failed induction courses.
3. Remission consolidation was risk-oriented, the risk being defined through a mixed clinico-cytogenetic model. Thus all patients entering CR after one/two cycles were stratified as HR or SR according to what is reported below. Once defined the risk class, therapy consisted of an alloSCT for HR patients, and of 3 consecutive monthly cytarabine-based cycles (2 g/m2/bd on days 1-5; idarubicin on days 1,2) in SR patients, each cycle being followed by the reinfusion of a limited amount of autologous blood stem cells (1-2x10e6/kg CD34+ cells) and G-CSF. Blood stem cells were collected following an early consolidation cycle with intermediate-dose cytarabine plus G-CSF. HR patients unable/unfit to proceed to alloSCT were offered instead the SR-type multicycle cytarabine consolidation, whereas all patients unable to mobilize autologous stem cells were treated with one/two intermediate-dose cytarabine course(s).

HR: high-risk cytogenetics or intermediate-risk/normal cytogenetics with FLT3 mutation and/or any one or more additional clinical risk factor(s), i.e. total WBC >50x10e9/l, FAB subtype M0, M6 or M7, prior myelodysplasia or secondary AML,hepatosplenomegaly, late CR (cycle 2), or favorable cytogenetics with late CR (cycle 2).

SR: favorable cytogenetics (without associated high-risk abnormalities and in CR after cycle 1) or intermediate-risk/normal cytogenetics without FLT3 mutation and/or without any one additional clinical risk factor(s), i.e. total WBC >50x10e9/l, FAB subtype M0, M6 or M7, prior myelodysplasia or secondary AML,hepatosplenomegaly, late CR (cycle 2).

ELIGIBILITY:
Inclusion Criteria:

* age 15-65 years,untreated AML (de novo, secondary, myelodysplasia-related, granulocytic sarcoma),untreated high-risk myelodysplasia (RAEB, RAEB-T), informed consent

Exclusion Criteria:

* acute promyelocytic leukemia, comorbidity precluding intensive chemotherapy approaches

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2000-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 5-years
  Percent of patients who are disease-free 5 years from start of therapy

SECONDARY OUTCOMES:
Complete remission | Two months
  Percent of patients who achieve complete remission within two months from start of therapy (i.e. after two chemotherapy cycles)
Overall survival | 5 years
  Percent of patients who are alive 5 years after diagnosis
Cumulative incidence of relapse | 5 years
  Percent of patients who suffer from leukemia relapse at 5 years from date of remission
Toxicity | 5 years
  Percent of patients who die of treatment-related complications (in different prognostic/treatment groups)until 5 years from start of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Renato Bassan, MD, Principal Investigator — Ospedali Riuniti di Bergamo USC Ematologia
Locations (12):
- Italy (12):
  - USC Ematologia Ospedali Riuniti di Bergamo, Bergamo, BG
  - Divisione Ematologia Spedali Civili di Brescia, Brescia, BS
  - Divisione di Ematologia e TMO Ospedale San Maurizio, Bolzano, BZ
  - Ematologia Azienda Ospedaliera S. Croce e Carle, Cuneo, CN
  - Ematologia e TMO Ospedale San Raffaele, Milan, MI
  - Ematologia e TMO Istituto Nazionale dei Tumori, Milan, MI
  - Ematologia-TMO Ospedale San Gerardo, Monza, MI
  - Oncoematologia e TMO Dipartimento Oncologico, Palermo, PA
  - Ematologia 2 Ospedale San Giovanni Battista, Torino, TO
  - Medicina Interna I Ospedale di Circolo, Varese, VA
  - Divisione Ematologia Ospedale Umberto I Mestre, Mestre, VE
  - Dipartimento di Oncologia e di Ematologia Oncologica Regione Veneto ULSS n.13- Presidi Ospedalieri di Noale, Dolo, Mirano, Noale, VE

REFERENCES:
- [Derived] Borlenghi E, Cattaneo C, Bertoli D, Cerqui E, Archetti S, Passi A, Oberti M, Zollner T, Giupponi C, Pagani C, Bianchetti N, Bottelli C, Bagnasco S, Sciume M, Tucci A, Rossi G. Prognostic Relevance of NPM1 and FLT3 Mutations in Acute Myeloid Leukaemia, Longterm Follow-Up-A Single Center Experience. Cancers (Basel). 2022 Sep 28;14(19):4716. doi: 10.3390/cancers14194716. PMID 36230640